CLINICAL TRIAL: NCT06699914
Title: A Retrospective, 12-month, Multicenter Study to Evaluate Real-world Brolucizumab Effectiveness and Safety in Japanese Patients With Neovascular Age-related Macular Degeneration (nAMD) - the PHEASANT Study - a Study Following the Master Protocol
Brief Title: A Study to Evaluate Real-world Brolucizumab Effectiveness and Safety in Japanese Patients With Neovascular Age-related Macular Degeneration (nAMD)
Acronym: PHEASANT
Status: Completed | Type: Observational
Sponsor: Novartis Pharmaceuticals (Industry)
Responsible Party: Sponsor
Organization: Novartis (Industry)
Other Study IDs: CRTH258A1001
Record Dates: First submitted 2024-11-19; First posted 2024-11-21 (Actual); Last update posted 2024-11-21 (Actual); Status verified 2024-11

CONDITIONS: Neovascular Age-Related Macular Degeneration

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective

GROUPS / COHORTS (2):
- Naive Group: Japanese patients diagnosed with nAMD who did not receive any anti-vascular endothelial growth factor (VEGF) injections during the 12 months before receiving brolucizumab.
- Pre-treated Group: Japanese patients diagnosed with nAMD who received at least one injection of another anti-VEGF treatment during the 12 months before receiving brolucizumab.

SUMMARY:
A retrospective, observational, single-arm, non-randomized cohort study of ocular treatment in nAMD patients in Japan who had records of at least 12 months of follow-up after their first brolucizumab intravitreal injection. Patients who had records of at least 12 months of visits after the first brolucizumab injection (index date) were identified during the index period and were recruited during the data collection/recruitment period.

ELIGIBILITY:
Inclusion criteria:

1. Diagnosis of nAMD.
2. Patients 50 years of age or older at index.
3. Received first injection of brolucizumab during the index period.
4. Gave signed or verbal informed consent.

Exclusion criteria:

1. Patients treated for retinal vein occlusion (RVO), diabetic macular edema (DME), myopic choroidal neovascularization (mCNV), and who had diagnoses of diabetes-related macular degeneration within 6 Months prior to the index date.
2. Any active intraocular or periocular infection or active intraocular inflammation in the study eye at index date.
3. Patients who had any contraindication and were not eligible for treatment with brolucizumab according to the label.
4. Patients who were treated with more than 3 types of anti-vascular endothelial growth factor (anti-VEGF) before the index date (5th line brolucizumab patients or more).
5. Patients participating in parallel in an interventional clinical trial.
6. Patients participating in post-marketing surveillance with brolucizumab.

Min Age: 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: This was a retrospective, noninterventional cohort study.
Sampling Method: Non-Probability Sample
Enrollment: 438 (Actual)
Dates: Start 2022-09-06 (Actual); Primary Completion 2023-12-01 (Actual); Study Completion 2023-12-01 (Actual)

PRIMARY OUTCOMES:
Number of Patients With Absence of Intra-retinal Fluid (IRF) and Absence of Subretinal Fluid (SRF) at Month 12 | Month 12
Number of Patients With Absence of IRF and Absence of SRF at Month 3, 6, 9, and 18 | Month 3, 6, 9, and 18

SECONDARY OUTCOMES:
Demographic: Age | Baseline
Demographic: Number of Patients per Age Category | Baseline
  Age categories:
  * Less than 80 years old.
  * 80 years or older.
Demographic: Gender | Baseline
Number of Patients per Clinical Characteristic | Baseline
  Clinical characteristics included:
  * Bilateral age-related macular degeneration (AMD)
  * Subtype of AMD, choroidal neovascularization (CNV)
  * CNV type (Type I, II, III, polypoidal choroidal vasculopathy (PCV) [yes/no/not graded])
  * Intra-retinal fluid (IRF)
  * Subretinal fluid (SRF)
  * Presence of SRF and/or IRF
  * Absence of SRF and IRF
  * Sub-retinal pigment epithelium (sub-RPE) fluid
Clinical Characteristic: Time Between Diagnosis and First Brolucizumab Injection | Baseline
Clinical Characteristic: Time Between Diagnosis and First Treatment | Baseline
Clinical Characteristic: Central Subfield Thickness (CSFT) | Baseline
Clinical Characteristic: Visual Acuity (VA) | Baseline
  Visual Acuity (VA) was measured with Early Treatment Diabetic Retinopathy Study (ETDRS) letters.
  Conversion of VA readings to approximate ETDRS Letters:
  * For Snellen fraction decimal >0.025 (<logMAR1.60) the following formula was used:
    • approximate ETDRS Letters = 85+50*log10 (Snellen fraction)
  * For Snellen fractions decimal ≤0.025 four bins were defined:
    * >0.020 to 0.025 (logMAR 1.70 to 1.60) was 5 letters
    * >0.015 to 0.020 (logMAR 1.82 to 1.70) was 3 letters
    * >0.005 to 0.015 (logMAR 2.30 to 1.82) was 1 letter
    * ≤0.005 (logMAR ≥2.30) is 0 letter
Clinical Characteristic: VA in Each Subtype | Baseline
  VA was measured with ETDRS letters. Subtypes included CNV Type I, II, III, PCV (yes/no/not graded).
Number of Patients by Type of Previous Anti-vascular Endothelial Growth Factor (Anti-VEGF) Treatment | Up to 12 months pre-baseline
Last Injection Interval of Anti-VEGF Treatment Before Switching | Up to 12 months pre-baseline
Number of Injections in the Last 6 Months Before Switching to Brolucizumab | Up to 6 months pre-baseline
Number of Injections in the Last 6 Months After Switching to Brolucizumab | Up to 6 months post-baseline
Number of Injections in the Last 12 Months Before Switching to Brolucizumab | Up to 12 months pre-baseline
Number of Injections in the Last 12 Months After Switching to Brolucizumab | Up to 12 months post-baseline
Number of Patients With Absence of Subretinal Fluid (SRF) | Month 3, 6, 9, 12 and 18
Number of Patients with Absence of Intra-retinal Fluid (IRF) | Month 3, 6, 9, 12, and 18
Number of Patients with Absence of Sub-retinal Pigment Epithelium (sub-RPE) Fluid | Month 3, 6, 9, 12, and 18
Number of Patients with Absence of SRF and IRF | Month 3, 6, 9, 12, and 18
Number of Patients with Absence of IRF, SRF, and sub-RPE Fluid | Month 3, 6, 9, 12, and 18
Time to Absence of Retinal Fluid During the First Year of Treatment Among Those With Presence of Retinal Fluid at Baseline | 12 months
  Retinal fluid categories included:
  * SRF
  * IRF
  * Sub-RPE
  * SRF and IRF
  * SRF, IRF, and sub-RPE
Central Subfield Thickness (CFST) at Month 3, 6, 9, 12 and 18 | Month 3, 6, 9, 12, and 18
Change in CFST From Baseline to Months 3, 6, 9, 12, and 18 | Baseline, Month 3, 6, 9, 12, and 18
VA Change in Each Subtype From Baseline to Month 3 | Baseline, Month 3
  VA was measured with ETDRS letters. Subtypes included CNV Type I, II, III, PCV (yes/no/not graded).
VA Change in Each Subtype From Baseline to Month 6 | Baseline, Month 6
  VA was measured with ETDRS letters. Subtypes included CNV Type I, II, III, PCV (yes/no/not graded).
VA Change in Each Subtype From Baseline to Month 9 | Baseline, Month 9
  VA was measured with ETDRS letters. Subtypes included CNV Type I, II, III, PCV (yes/no/not graded).
VA Change in Each Subtype From Baseline to Month 12 | Baseline, Month 12
  VA was measured with ETDRS letters. Subtypes included CNV Type I, II, III, PCV (yes/no/not graded).
VA Change in Each Subtype From Baseline to Month 18 | Baseline, Month 18
  VA was measured with ETDRS letters. Subtypes included CNV Type I, II, III, PCV (yes/no/not graded).
Number of Brolucizumab Injections During the Study Within Specified Time Intervals | Up to 18 months
  Time intervals included:
  * 0 to 3 months
  * 3 to 6 months
  * 6 to 12 months
  * 13 to 18 months
  * 0 to 12 months
  * 0 to 18 months
Number of Non-injection Visits During Treatment With Brolucizumab Within Specified Time Intervals | Up to 18 months
  Time intervals included:
  * 0 to 3 months
  * 3 to 6 months
  * 6 to 12 months
  * 13 to 18 months
  * 0 to 12 months
  * 0 to 18 months
Number of Visits During Treatment With Brolucizumab Within Specified Time Intervals | Up to 18 months
  Time intervals included:
  * 0 to 3 months
  * 3 to 6 months
  * 6 to 12 months
  * 13 to 18 months
  * 0 to 12 months
  * 0 to 18 months
Number of Patients Categorized by Injection Intervals During Months 0 to 6 | From Month 0 to Month 6
  Injection intervals (weeks) included:
  * Less than 4 weeks
  * ≥4 weeks but <6 weeks
  * ≥6 weeks but <8 weeks
  * ≥8 weeks but <10 weeks
  * ≥10 weeks but <12 weeks
  * ≥12 weeks but <14 weeks
  * ≥14 weeks but <16 weeks
  * ≥16 weeks but <20 weeks
  * 12 weeks or more
  * 16 weeks or more
  * 20 weeks or more
Number of Patients Categorized by Injection Intervals During Months 0 to 12 | From Month 0 to Month 12
  Injection intervals (weeks) included:
  * Less than 4 weeks
  * ≥4 weeks but <6 weeks
  * ≥6 weeks but <8 weeks
  * ≥8 weeks but <10 weeks
  * ≥10 weeks but <12 weeks
  * ≥12 weeks but <14 weeks
  * ≥14 weeks but <16 weeks
  * ≥16 weeks but <20 weeks
  * 12 weeks or more
  * 16 weeks or more
  * 20 weeks or more
Number of Patients Categorized by Injection Intervals During Months 0 to 18 | From Month 0 to Month 18
  Injection intervals (weeks) included:
  * Less than 4 weeks
  * ≥4 weeks but <6 weeks
  * ≥6 weeks but <8 weeks
  * ≥8 weeks but <10 weeks
  * ≥10 weeks but <12 weeks
  * ≥12 weeks but <14 weeks
  * ≥14 weeks but <16 weeks
  * ≥16 weeks but <20 weeks
  * 12 weeks or more
  * 16 weeks or more
  * 20 weeks or more
Number of Patients Categorized by Injection Intervals During Months 13 to 18 | From Month 13 to Month 18
  Injection intervals (weeks) included:
  * Less than 4 weeks
  * ≥4 weeks but <6 weeks
  * ≥6 weeks but <8 weeks
  * ≥8 weeks but <10 weeks
  * ≥10 weeks but <12 weeks
  * ≥12 weeks but <14 weeks
  * ≥14 weeks but <16 weeks
  * ≥16 weeks but <20 weeks
  * 12 weeks or more
  * 16 weeks or more
  * 20 weeks or more
Number of Patients With a Change in Injection Interval at Month 12 | Month 12
  Changes in injection interval included:
  * Prolonged (1 week or more)
  * Stable
  * Reduced (1 week or less)
Number of Patients With Prophylactic Administration of Steroid Eye Drops Within Specified Time Intervals | Up to 18 months
  Time intervals included:
  * Month 0 to 3
  * Month 3 to 6
  * Month 6 to 12
  * Month 13 to 18
Number of Visits With Optical Coherence Tomography (OCT) Within Specified Time Intervals | Up to 18 months
  Time intervals included:
  * 0 to 6 months
  * 0 to 12 months
  * 0 to 18 months
  * 13 to 18 months
Number of Visits Without OCT Within Specified Time Intervals | Up to 18 months
  Time intervals included:
  * 0 to 6 months
  * 0 to 12 months
  * 0 to 18 months
  * 13 to 18 months
Predictive Variables of VA Change From Baseline to Month 12 | Baseline, Month 12
  A multivariate regression model was used to assess the predictive value of VA change from baseline. Independent variables included age, baseline VA, baseline CNV activity, loading phase, VA (ETDRS letters) at the end of loading phase, CNV activity at the end of loading phase, PCV activity, number of injections, and geographic atrophy.
Number of Patients Categorized by Criteria for Re-treatment | Month 3, 6, 9, 12, and 18
  Re-treatment criteria included VA, anatomic parameters, VA and anatomic parameters, and posology requirement.
Number of Patients Categorized by Criteria for No Re-treatment | Month 3, 6, 9, 12, and 18
  No re-treatment criteria included general visits and check of brolucizumab related intraocular inflammation (IOI).
Number of Patients who Switched to Another Anti-VEGF During Treatment With Brolucizumab Within Specified Time Intervals | Up to 18 months
  Time intervals included:
  * Month 0 to 3
  * Month 3 to 6
  * Month 6 to 9
  * Month 9 to 12
  * After 12 months
Number of Patients who Discontinued Treatment During the First Year | Up to 12 months
Number of Patients by Reason for Discontinuing Brolucizumab Treatment | Up to 12 months
Number of Patients With Adverse Events (AEs) | Up to 12 months
Number of Patients With Adverse Events of Special Interest (AESIs) and by Type of AESI | Up to 12 months
  AESIs included endophthalmitis and Intraocular inflammation (IOI) including vasculitis and retinal vascular occlusion.
Number of AEs and AESIs per Patients | Up to 12 months
Number of Patients With AEs Categorized by Age and Gender | Up to 12 months
Number of Patients With AESIs Categorized by Age and Gender | Up to 12 months
Number of Patients With Brolucizumab-related AEs and AESIs | Up to 12 months
Number or Patients Who's AEs and AESIs Resolved | Up to 12 months
Number of Resolved AEs and AESIs | Up to 12 months
Time From First Brolucizumab Injection to AESIs | Up to 12 months
Best Corrected Visual Acuity (BCVA) | Up to 12 months
  BCVA was assessed before AESI onset, during AESI, and after AESI recovery. BCVA is the best possible vision that an eye can achieve with the use of glasses or contact lenses. It is measured by ETDRS chart or Snellen chart.

CONTACTS AND LOCATIONS:
Overall Officials: Novartis Pharmaceuticals, Study Director — Novartis Pharmaceuticals
Locations (1):
- Novartis, East Hanover, New Jersey, United States

REFERENCES:
- [Derived] Ohnaka M, Sakurada Y, Hayashi A, Kadonosono K, Ohno H, Mori R, Matsumoto H, Nagamori I, Murata Y, Maio-Twofoot T, Karcher H, Takahashi H. Real-World Outcomes of Brolucizumab Treatment in Japanese Patients with Neovascular Age-Related Macular Degeneration: A 12-Month, Multicenter Study. Ophthalmol Ther. 2025 Jul;14(7):1551-1565. doi: 10.1007/s40123-025-01159-2. Epub 2025 May 28. PMID 40434532